CLINICAL TRIAL: NCT01968863
Title: Evaluation of a Microendoscopic Imaging System in Examination of Resected Tissues
Status: Terminated | Type: Observational
Why Stopped: Investigator Non Compliance
Sponsor: University of Arkansas (Other)
Collaborators: University of Arkansas, Fayetteville (Other)
Responsible Party: Sponsor
Other Study IDs: 202224
Record Dates: First submitted 2013-10-15; First posted 2013-10-24 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Known or Suspected Dysplasia or Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall objective of this exploratory, laboratory study is to evaluate whether noninvasive fluorescence microendoscopic imaging of tissue can assist clinicians in detecting dysplastic (precancerous) areas during standard surveillance. This is a study designed to evaluate the feasibility of using prototype imaging technology to enhance the detection of precancerous changes in various tissues. The results of this laboratory study will be used to further develop the technology for clinical application.

The primary aim of this project will be to investigate what digital image analysis criteria can be used to best detect dysplasia in various types of resected tissue.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over the age of 18 scheduled for standard of care resection of abnormal tissue

Exclusion Criteria:

* Previous chemotherapy or radiation treatment to the tissue to be resected
* Inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with known or suspected dysplasia or cancer scheduled to undergo either endoscopic or surgical resection will be approached for participation.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Statistical measurements of the spatial and intensity distributions of pixels within an image | Up to 24 hours
  The statistical measurements will be used to correlate each microendoscope image to a histopathology diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States